CLINICAL TRIAL: NCT06320015
Title: Emergency Department Community Health Worker-Peer Recovery Navigation for Linkage to Recovery: A Mixed Methods Evaluation
Brief Title: Emergency Medicine Peer Outreach Worker Engagement for Recovery
Acronym: EMPOWER
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Brown University (Other)
Responsible Party: Principal Investigator, Elizabeth Samuels, Associate Professor, University of California, Los Angeles
Other Study IDs: R01CE003632-01-00; R01CE003632 (NIH)
Record Dates: First submitted 2023-11-18; First posted 2024-03-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorders; Overdose; Opioid Use Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Substance-Related Disorders; Drug Overdose; Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SMART Participant: Emergency department patients at with a substance use disorder who have received SMART services
  Interventions: Behavioral: Substance Misuse Assistance Response Team (SMART)
- Usual Care: Emergency department patients with a substance use disorder who have not received SMART services
  Interventions: Other: Usual Care Group

INTERVENTIONS:
Behavioral: Substance Misuse Assistance Response Team (SMART) — The study intervention is engagement with a Substance Misuse Assistance Response Team (SMART) community health worker-peer recovery specialist (PCHW). SMART PCHWs engage ED patients with substance use disorders and facilitates ED services provision and linkages to outpatient care. Services provided include supporting ED initiation of buprenorphine, harm reduction services, social services (transportation, housing assistance, etc.), and engagement in peer recovery, behavioral health services, and addiction treatment services. Services are provided at the time of the ED visit. A subgroup of patients is provided short term case management and outpatient services navigation depending on PCHW caseload availability and individual needs.
  Groups: SMART Participant
Other: Usual Care Group — Patient not seen by a SMART community health worker in the emergency department. Care and treatment referral at discretion of emergency department treating team.
  Groups: Usual Care

SUMMARY:
This is an observational, prospective case-control study evaluating the effects of an emergency department community health worker-peer recovery specialist program (PCHW), the Substance Misuse Assistance Response Team (SMART). Aims of this study are to 1) understand participant experiences working with a SMART PCHW and identify possible mechanisms for successful recovery linkage; 2) Evaluate SMART effectiveness on patient-centered outcomes, building recovery capital, and recovery linkage; 3) Evaluate SMART implementation and effectiveness on patient outcomes over time.

Using a combination of surveys and data linkages to state administrative databases, study investigators will prospectively compare changes in addiction treatment engagement, recovery capital, health related social needs, acute care utilization, and death between people receiving a ED PCHW and those who do not. After consenting to study participation, participants will complete surveys at time of study enrollment and 3 and 6 months after their initial ED visit. Primary outcomes include engagement in addiction treatment, social services engagement, acute care utilization, and mortality will be assessed through linkages to state administrative databases.

DETAILED DESCRIPTION:
The emergency department (ED) is on the front lines of the overdose epidemic, treating an increasing number of people with substance use disorders (SUD). In the year after a substance use-related ED visit, risk of death is six time higher than other patients, and for people treated after an opioid overdose, more than one in twenty patients will die. Each substance use-related ED visit represents a crucial opportunity to link patients to recovery services, however there are significant gaps in service provision with less than one in three receiving behavioral counseling and only one in five linked to addiction treatment. To improve linkage to recovery and addiction treatment services from the ED, study investigators launched a multidisciplinary, ED community health worker-peer recovery specialist program (PCHW), the Substance Misuse Assistance Response Team (SMART), at a large, academic, urban medical center which cares for the majority of patients with SUDs in Rhode Island. Drawing from models of existing peer recovery specialist, CHW, and health promotion advocate programs, SMART is a novel ED-based program that provides people with a substance-use related ED visit individualized support, short term case management, navigation to social services, harm reduction, recovery, and addiction treatment services in and out of the ED. SMART distinguishes itself from other models of ED patient navigation and/or peer recovery specialist programs by working in and out of the ED and focusing on social determinants of recovery. In recent years there has been a proliferation of ED peer recovery programs, but little is known about their effectiveness. Study investigators will conduct a pragmatic, mixed methods study of an established ED PCHW program to evaluate program delivery, linkage to evidence-based recovery services, and short- and long-term patient outcomes. Aims of this study are to 1) understand participant experiences working with a SMART PCHW and identify possible mechanisms for successful recovery linkage; 2) Evaluate SMART effectiveness on patient-centered outcomes, building recovery capital, and recovery linkage; 3) Evaluate SMART implementation and effectiveness on patient outcomes over time. Participant interviews will examine participant experiences with SMART, recovery services engagement, and identify potentially effective engagement strategies. A RE-AIM framework will be used to evaluate program implementation (process outcomes) and effectiveness (patient outcomes). Surveys and data linkage to hospital and state administrative databases will be used to measure changes in recovery capital, social networks, receipt of social services, linkage to harm reduction, recovery, and addiction treatment services, and changes in acute care utilization and mortality among people receiving SMART. Results from this study will provide robust data about ED peer recovery specialist program process and patient-level outcomes needed for a subsequent multilevel, comprehensive study to identify and test effectiveness of ED peer recovery program components and implementation strategies for program enhancement, dissemination, and sustainability.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years old or older
2. Seen and treated at Rhode Island or The Miriam Hospital ED for a substance use-related concern including intoxication, withdrawal, opioid overdose, opioid withdrawal, or substance use-related infection
3. Able to provide informed consent
4. Able to provide at least two forms of contact (personal phone, social media, email, or contact information for family or friends)
5. Participants may speak languages other than English but require use of interpreter services. Consents will be available in English, Spanish, and Portuguese, the three most spoken languages in the Providence metropolitan area.

Exclusion Criteria:

1. Unable to provide informed consent
2. In police custody, incarcerated, or have a court ordered treatment enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll 400 people with a substance-used related visit. Individuals will be approached after receipt of ED services.
  1. 200 people who have received SMART services.
     - Participants will be approached for study participation after they have already received SMART services.
  2. 200 people who did NOT receive SMART services.
     * Participants will be approached for study enrollment in this study arm when they are seen and treated on a day and time or ED site where SMART is not available.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Treatment engagement | Will compare differences in treatment engagement between study arms 3 and 6 months after study enrollment.
  Investigators will measure engagement in formal addiction treatment at a state licensed addiction treatment facility and/or receipt of office-based buprenorphine through data linkages to the Rhode Island Prescription Drug Monitoring Program database and the Rhode Island Behavioral Health Online Database.
Recovery Capital | Will compare differences in treatment engagement between study arms 3 and 6 months after study enrollment.
  Investigators will conduct surveys with study participants at time of enrollment, three months after enrollment, and six months after enrollment. Survey Changes in individual recovery capital as measured by reported self-efficacy, social networks, and quality of life

SECONDARY OUTCOMES:
Emergency Department Utilization | Will compare differences in acute care utilization between study arms 3 and 6 months after study enrollment.
  Investigators will measure emergency department utilization through review of health system electronic health records and data linkages to the Rhode Island Emergency Medical Services and Medicaid claims databases.
Repeat Hospitalization | Will compare differences in acute care utilization between study arms 3 and 6 months after study enrollment.
  Investigators will measure hospitalizations review of health system electronic health records and data linkages to the Rhode Island Emergency Medical Services and Medicaid claims databases.
Repeat Overdose | Will compare differences in acute care utilization between study arms 3 and 6 months after study enrollment.
  Investigators will measure overdose incidence review of health system electronic health records and data linkages to the Rhode Island Emergency Medical Services and Medicaid claims databases.
Mortality | Will compare differences in mortality between study arms 3 and 6 months after study enrollment.
  Through linkage to the state vital records database, investigators will compare differences in mortality between study arms.
Social Services Engagement | Will compare differences in health related social needs between study arms 3 and 6 months after study enrollment.
  Investigators will compare changes in social services engagement needs through linkage to the Rhode Island Executive Office of Health and Human Services Data Ecosystem. Databases included in the Data Ecosystem include the Rhode Island Department of Labor and Training, Department of Health and Human Services, Department of Corrections, Department of Human Services, and the Rhode Island Coalition on Homelessness.
Housing Services Engagement | Will compare differences in housing services engagement between study arms 3 and 6 months after study enrollment.
  Investigators will compare changes in housing services engagement for participants unstably housed. Participants will be identified as unstably housed through study intake survey responses. Outcomes will be identified through linkage to the Rhode Island Coalition on Homelessness data housed in the Rhode Island Executive Office of Health and Human Services Data Ecosystem.
Employment | compare differences in changes in employment between study arms 3 and 6 months after study enrollment.
  Investigators will compare changes in employment through linkage to the Rhode Island Department of Labor and Training databased housed in the Rhode Island Executive Office of Health and Human Services Data Ecosystem.
Incarceration | Will compare differences in changes in incarceration and encounters with the criminal justice system between study arms 3 and 6 months after study enrollment.
  Investigators will compare changes in incarceration and encounters with the criminal justice system through linkage to the Rhode Island Department of Corrections database which is housed in the Rhode Island Executive Office of Health and Human Services Data Ecosystem.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Samuels, MD, MPH, MHS, Principal Investigator — UCLA Emergency Medicine
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No